CLINICAL TRIAL: NCT03563651
Title: A Pilot Study of Monitoring Metastatic Colorectal Cancers With Liquid Biopsies
Brief Title: Collection of Blood, Urine, and Stool to Monitor MetastaticColorectal Cancers
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 3C-13-2; NCI-2018-00801 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 3C-13-2 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2018-06-09; First posted 2018-06-20 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Stage III Colorectal Cancer AJCC v8; Stage IIIA Colorectal Cancer AJCC v8; Stage IIIB Colorectal Cancer AJCC v8; Stage IIIC Colorectal Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, stool
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (biospecimen collection, biopsy): Participants undergo collection of blood and urine at baseline, on day 1 of courses 1, 2, and 3, at restaging, and at disease progression. Participants may undergo collection of stool at baseline, on day 1 of course 2, and at disease progression. Participants also undergo biopsy within 4 weeks of disease progression.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: Bx
Procedure: Biospecimen Collection — Undergo collection of blood, urine, and stool
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies the monitoring of therapy and progression by collecting blood, urine, and stool from participants with colorectal cancer that has spread to other places in the body or cannot be removed by surgery. Studying samples of blood, urine, and stool from participants with colorectal cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Detection of mutated Kras in urine specimen of patients with Kras mutated metastatic colon cancer on first, second, or third line therapy.

II. Detection of new Kras in urine in patients without Kras mutated metastatic colon cancer on therapy which includes anti-EGFR antibodies (cetuximab or panitumumab).

SECONDARY OBJECTIVES:

I. Changes of the stool microbiome with chemotherapy and at progression of the disease.

DESCRIPTIVE OBJECTIVES:

I. Changes in the quantity of mutated Kras, Braf or PI3K in urine deoxyribonucleic acid (DNA) over the cycles of first line therapy.

II. Associations between the quantity of mutated Kras, Braf or PI3K in urine DNA, molecular make up of circulating tumor cells (CTCs), cell free DNA and progression over the course of first line therapy.

III. Feasibility of detection of exosome in the plasma of colorectal cancer patients on first line chemotherapy in Dr. Fabbri?s lab at Children?s Hospital Los Angeles.

IV. Feasibility of detection of tumor DNA in the plasma of colorectal cancer patients on first line chemotherapy.

OUTLINE:

Participants undergo collection of blood and urine at baseline, on day 1 of courses 1, 2, and 3, at restaging, and at disease progression. Participants may undergo collection of stool at baseline, on day 1 of course 2, and at disease progression. Participants also undergo biopsy within 4 weeks of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* All patients with metastatic/unresectable colorectal cancer who will undergo first, second, or third line therapy; the participating investigator will select treatment, however, patients with Kras wild type must receive anti-EGFR therapy to be eligible for this study
* Subject consent to enrollment on the protocol
* Histologically confirmed metastatic or un-resectable colorectal cancer, known Kras status; knowledge of other mutations is optional
* Willingness to undergo biopsy at the time of progression
* Willingness to follow the study instructions for collection of specimens
* Available archival tissue

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with metastatic/unresectable colorectal cancer who will undergo first, second, or third line therapy at USC facilities will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2014-02-06 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
Detection rates of Kras, Braf, or PI3K tumor deoxyribonucleic acid (DNA) extracted from urine in patients with pre-existing mutations | Up to 5 years
  Mutation detection rate will be estimated by gene and treatment cycle in each cohort. The quantities of mutated Kras, Braf, or PI3K will be estimated using means and standard deviation if the distribution of the quantities is compatible with normal distribution. Otherwise, medians, ranges and interquartiles will be used. The changes in the mutation status and quantities of Kras, Braf, and PI3K before and after starting the first line therapy will be estimated using contingency tables and plots.
Detection rates of Kras, Braf, or PI3K tumor DNA extracted from urine in patients without pre-existing mutations | Up to 5 years
  Mutation detection rate will be estimated by gene and treatment cycle in each cohort. The quantities of mutated Kras, Braf, or PI3K will be estimated using means and standard deviation if the distribution of the quantities is compatible with normal distribution. Otherwise, medians, ranges and interquartiles will be used. The changes in the mutation status and quantities of Kras, Braf, and PI3K before and after starting the first line therapy will be estimated using contingency tables and plots.

CONTACTS AND LOCATIONS:
Overall Officials: Afsaneh Barzi, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States